

## INFORMED CONSENT FOR THE PATIENT

Correlation of pupillary diameter change with age and anterior chamber depth after cataract surgery

Approved by the CEIm Grupo Hospitalario Quirónsalud-Catalunya on June 21, 2018 (ID: 47/2018)



## **INFORMED CONSENT FOR THE PATIENT**

## STUDY EC022018

Correlation of the change in pupillary diameter with age and anterior chamber depth after cataract surgery

| l, | |
|---|---|
| (patient's full name) | |
| I have read the information sheet g | given to me |
| I have been able to ask questions a | _ |
| I have received enough information | • |
| I have been informed by the resear | • |
| <ul> <li>I understand that my part<br/>collected in the conditions detailed</li> </ul> | ticipation is voluntary and that the data will be d in the Patient Information Sheet. |
| of Personal Data, the consent for t | nish Law 15/1999 of December 13, on the Protection he processing of your personal data and for its cise the right of access, rectification and cancellation |
| o Without having to | ithdraw from the study or anytime. give explanations. ng an impact on my care in the study. |
| o without this havin | is an impact on my care in the study. |
| <ul> <li>I freely give my agreemen</li> </ul> | nt to participate in the study. |
| Patient Signature | Investigator Signature |
| Name: | Name: |

Date:

Date: